CLINICAL TRIAL: NCT02499302
Title: Mental Training for Chronic Fatigue Syndrome (CFS/ME) Following EBV Infection in Adolescents: A Randomised Controlled Trial
Brief Title: Mental Training for CFS Following EBV Infection in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Wyller, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBA part 2
Record Dates: First submitted 2015-07-09; First posted 2015-07-16 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Fatigue Syndrome, Chronic; Epstein-Barr Virus Infection
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Epstein-Barr Virus Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mental training (Experimental): The intervention consists of one introductory session (patients and their parents/next-of-kin), followed by 9 individual therapy sessions (one each week) of 1.5 hours duration and related home-work, combining elements from cognitive behavioural therapy and music therapy: Important elements of the mental training program are:
  * Psychoeducation: Theories of CFS/ME pathophysiology and treatment rationale
  * Relaxation: Bodily stress reduction, mindfulness
  * Visualization: Contact with positive emotions, techniques of worrying reduction
  * Experiences: Behavioral 'experiments' (individually adjusted), 'trick into action'
  * Cognitive challenges: Challenging thoughts about disease process, stimulus and outcome expectancies, prognosis
  Interventions: Behavioral: Mental training
- Routine follow-up (No Intervention): Routine follow-up by the general practitioner, which is normal approach to chronic fatigue following acute EBV infection.

INTERVENTIONS:
Behavioral: Mental training
  Arms: Mental training

SUMMARY:
The general aim of this study is to investigate the effect of an individually tailored mental training program in adolescents developing chronic fatigue syndrome (CFS) after an acute Epstein Barr-virus (EBV) infection. Endpoints include physical activity (primary endpoint), symptoms (fatigue, pain, insomnia), cognitive function (executive functions) and markers of disease mechanisms (autonomic, endocrine, and immune responses).

DETAILED DESCRIPTION:
EBV-infection is a well-known trigger of CFS. A closely related research project (Chronic fatigue following acute Epstein-Barr virus infection in Adolescents; ClinicalTrials ID:NCT02335437) is a combined prospective and cross-sectional study of 200 adolescents suffering from acute EBV infection. The primary aim of that study is to identify factors that predispose to CFS 6 months after the acute infection. Thus, that project will provide a sample of thoroughly characterized CFS patients, all having the same precipitation factor (EBV-infection).

The present project is an intervention trial in the subgroup of patients that actually did develop CFS 6 months after the acute EBV infection. Patients will be randomised 1:1 to either a mental training program (10 sessions) combining elements from cognitive behavioral therapy and music therapy, or routine follow-up from the general practitioner. By its nature, treatment group allocation cannot be blinded; however, both patients and therapists will be blinded for end-point evaluation. An extensive investigational program will be carried out at three time points: Prior to the intervention, immediately after the intervention, and 1 year after the intervention. The program includes: Clinical examination; Pain threshold assessment; Cardiovascular assessment; Cognitive assessment; Sampling of biological material (blood and urine); Questionnaire; Brain fMRI; Qualitative interview; Monitoring of physical activity (accelerometer)

ELIGIBILITY:
Inclusion Criteria:

* Participant in the research project CEBA (Chronic fatigue following acute Epstein-Barr virus infection in adolescents, NCT02335437)
* Chronic fatigue at 6 months (a sum score of dichotomized responses ≥ 4 on the Chalder Fatigue questionnaire)

Exclusion Criteria:

* Other illnesses that might explain the fatigue
* Bedridden

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Physical activity | 12 weeks
  Mean steps/day during 7 consecutive days measured by accelerometer

SECONDARY OUTCOMES:
Plasma catecholamines | 12 weeks
Plasma catecholamines | 64 weeks
Urine cortisol:creatinin ratio | 12 weeks
Urine cortisol:creatinin ratio | 64 weeks
Degree centrality index of cytokine network | 12 weeks
  An index of node centrality, based upon network analyses
Degree centrality index of cytokine network | 64 weeks
  An index of node centrality, based upon network analyses
Number of NK-cells | 12 weeks
Number of NK-cells | 64 weeks
Supine heart rate | 12 weeks
Supine heart rate | 64 weeks
Heart rate variability indices | 12 weeks
Heart rate variability indices | 64 weeks
Heart rate, blood pressure and total peripheral resistence responses to upright posture | 12 weeks
Heart rate, blood pressure and total peripheral resistence responses to upright posture | 64 weeks
Working memory | 12 weeks
  Digit span forward and backward test
Working memory | 64 weeks
  Digit span forward and backward test
Cognitive inhibition | 12 weeks
  Color-word interference test from the D-KEFS instrument
Cognitive inhibition | 64 weeks
  Color-word interference test from the D-KEFS instrument
Correlation matrix indices of regions of interests (ROIs) in the brain salience network | 12 weeks
  Functional connectivity analyses from resting state brain fMRI
Correlation matrix indices of regions of interests (ROIs) in the brain salience network | 64 weeks
  Functional connectivity analyses from resting state brain fMRI
Fatigue score (Chalder fatigue questionnaire) | 12 weeks
Fatigue score (Chalder fatigue questionnaire) | 64 weeks
Pain scores (Brief pain Inventory) | 12 weeks
Pain scores (Brief pain Inventory) | 64 weeks
Quality of Life score (PedsQL) | 12 weeks
Quality of Life score (PedsQL) | 64 weeks
Anxiety and depression score (HADS) | 12 weeks
Anxiety and depression score (HADS) | 64 weeks
Alexithymia score (TAS-20) | 12 weeks
Alexithymia score (TAS-20) | 64 weeks
Insomnia score (KSQ) | 12 weeks
Insomnia score (KSQ) | 64 weeks
Pain threshold (algometry) | 12 weeks
Pain threshold (algometry) | 64 weeks
Disability score (FDI) | 12 weeks
Disability score (FDI) | 64 weeks
Side effect and unexpected events questionnaire | 3 weeks
Side effect and unexpected events questionnaire | 6 weeks
Side effect and unexpected events questionnaire | 9 weeks
Side effect and unexpected events questionnaire | 12 weeks
Physical activity | 64 weeks
  Mean steps/day during 7 consecutive days measured by accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Bruun Wyller, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Dept. of Pediatrics, Akershus University Hospital, Lørenskog, Akershus, Norway

REFERENCES:
- [Derived] Malik S, Asprusten TT, Pedersen M, Mangersnes J, Trondalen G, van Roy B, Skovlund E, Wyller VB. Cognitive-behavioural therapy combined with music therapy for chronic fatigue following Epstein-Barr virus infection in adolescents: a randomised controlled trial. BMJ Paediatr Open. 2020 Oct 21;4(1):e000797. doi: 10.1136/bmjpo-2020-000797. eCollection 2020. PMID 33117895
- [Derived] Malik S, Asprusten TT, Pedersen M, Mangersnes J, Trondalen G, van Roy B, Skovlund E, Wyller VB. Cognitive-behavioural therapy combined with music therapy for chronic fatigue following Epstein-Barr virus infection in adolescents: a feasibility study. BMJ Paediatr Open. 2020 Apr 9;4(1):e000620. doi: 10.1136/bmjpo-2019-000620. eCollection 2020. PMID 32342016 (Retraction: PMID 33123631 BMJ Paediatr Open. 2020 Oct 21;4(1):e000620ret)